CLINICAL TRIAL: NCT06122935
Title: Evaluation of the Aurora Xi New Nomogram Software 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenwal, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PAND-004-CMD
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Apheresis Related Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Test Group (Experimental): Plasma collection using a new plasma collection volume nomogram (software version 2.0) for the Aurora Xi Plasmapheresis System
  Interventions: Device: Aurora Xi New Nomogram Software 2.0
- Control Group (Active Comparator): Plasma collection using the marketed (version 1.3) of AuroraXi Plasmapheresis System
  Interventions: Device: Aurora Xi Currently Approved Software 1.3

INTERVENTIONS:
Device: Aurora Xi New Nomogram Software 2.0 — Plasma collection with a proprietary plasma collection volume nomogram provides a more individualized approach to determining the volume of plasma collected from each donor.
  Arms: Test Group
Device: Aurora Xi Currently Approved Software 1.3 — Plasma collection using the currently marketed Optimized Nomogram (software version 1.3) for the Aurora Xi Plasmapheresis System
  Arms: Control Group

SUMMARY:
A clinical trial to evaluate the safety and effectiveness of the Aurora Xi Plasmapheresis System with a new plasma collection volume nomogram.

DETAILED DESCRIPTION:
A controlled, prospective, randomized, multicenter, IDE clinical trial to evaluate the safety and effectiveness of a new plasma collection volume nomogram on the Aurora Xi Plasmapheresis System (test arm) as compared to the currently marketed Optimized Nomogram on the Aurora Xi Plasmapheresis System (control arm). The new plasma collection volume nomogram will provide a more individualized approach to determining the volume of plasma collected from each donor. The trial will be conducted at a minimum of 3 plasma collection centers. Subjects will be randomized into the test and control arms.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must meet current safety guidelines for plasma donation as set forth by the FDA as well as those in the standard operating procedures established by the participating institution.
* Enrolled subjects who do not meet inclusion criteria at a later donation attempt are eligible to remain in the clinical trial and to subsequently donate plasma once they meet eligibility criteria again.

Exclusion Criteria:

* Subjects not able or unwilling to give consent to participate.
* Subjects withdrawn by a qualified healthcare provider due to safety concerns.
* Subjects who are employed by the clinical site or Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6735 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Pineda, Study Director — Fresenius Kabi
Locations (3):
- United States (3):
  - BioLife Plasma Services, Lakeland, Florida
  - BioLife Plasma Services, West Des Moines, Iowa
  - BioLife Plasma Services, American Fork, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6,735 subjects were enrolled in the study at 3 investigative sites and completed 52,468 Per Protocol procedures.
Units Other Than Participants: Procedures
Period: Overall Study
Arm/Group | Test Group | Control Group
Started | 3363; 26351 Procedures | 3372; 26117 Procedures
Completed | 3363; 26351 Procedures | 3372; 26117 Procedures
Not Completed | 0; 0 Procedures | 0; 0 Procedures

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Group | Control Group | Total
Number analyzed (Participants) | 3363 | 3372 | 6735
Age, Customized [Mean (Standard Deviation); unit: years] | 36.9 (12.38) | 36.5 (12.53) | 36.7 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1521 | 1526 | 3047
  Male | 1842 | 1846 | 3688
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 630 | 642 | 1272
  Not Hispanic or Latino | 2704 | 2710 | 5414
  Unknown or Not Reported | 29 | 20 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 28 | 17 | 45
  Asian | 46 | 38 | 84
  Native Hawaiian or Other Pacific Islander | 39 | 35 | 74
  Black or African American | 275 | 272 | 547
  White | 2831 | 2853 | 5684
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 144 | 157 | 301
Region of Enrollment [Number; unit: participants]
  United States | 3363 | 3372 | 6735

OUTCOME MEASURES:

1. Primary Outcome: Rate of Significant Hypotensive Adverse Events
Description: The primary objective of this study is to demonstrate that the overall rate of significant hypotensive adverse events (SHAEs, IQPP DAE Classification 1.2-1.6) in donors using the Aurora Xi New Nomogram algorithm is less than double the SHAE rate in donors using the Aurora Xi Optimized Nomogram algorithm.
Time Frame: From venipuncture through 72 hours post-donation.
Measure: Number; unit: Procedure with a SHAE
Units Other Than Participants: Procedures
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 3363 | 3372
Number analyzed (Procedures) | 26351 | 26117
Procedure with a SHAE | 43 | 42

2. Secondary Outcome: Rate of Severe Hypotensive Adverse Events Relative to Donor Type
Description: To determine if the incidence rate of SHAEs per donor status (first-time donor) observed with the New Nomogram (Test arm) is non-inferior to the incidence rate observed with the Optimized Nomogram (Control arm).
Time Frame: From Venipuncture through 72 Hours post-donation.
Measure: Number; unit: Number of Participants with a SHAE
Units Other Than Participants: Procedures
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 1038 | 1043
Number analyzed (Procedures) | 1038 | 1043
Number of Participants with a SHAE | 9 | 5

3. Secondary Outcome: Rate of Severe Hypotensive Adverse Events Relative to Sex
Description: To determine if the incidence rate of SHAEs for female donors observed with the New Nomogram (Test arm) is non-inferior to the incidence rate observed with the Optimized Nomogram (Control arm).
Time Frame: From venipuncture through 72 hours post-donation.
Measure: Number; unit: Procedure with a SHAE
Units Other Than Participants: Procedures
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 1529 | 1532
Number analyzed (Procedures) | 11377 | 11372
Procedure with a SHAE | 31 | 29

4. Secondary Outcome: Rate of Severe Hypotensive Adverse Events Relative to Age
Description: To determine if the incidence rate of SHAEs for donors ≤20 years of age observed with the New Nomogram (Test arm) is non-inferior to the incidence rate observed with the Optimized Nomogram (Control arm).
Time Frame: From venipuncture through 72 hours post-donation.
Measure: Number; unit: Procedure with a SHAE
Units Other Than Participants: Procedures
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 229 | 250
Number analyzed (Procedures) | 1292 | 1452
Procedure with a SHAE | 5 | 5

5. Secondary Outcome: Rate of Severe Hypotensive Adverse Events Relative to Weight
Description: To determine if the incidence rate of SHAEs for donors weighting ≤124 lbs observed with the New Nomogram (Test arm) is non-inferior to the incidence rate observed with the Optimized Nomogram (Control arm).
Time Frame: From venipuncture through 72 hours post-donation.
Measure: Number; unit: Procedure with a SHAE
Units Other Than Participants: Procedures
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 75 | 81
Number analyzed (Procedures) | 476 | 465
Procedure with a SHAE | 1 | 2

6. Secondary Outcome: Rate of Hypotensive Severe/Injury Adverse Events (IQPP DAE Classification 1.5 or 1.6)
Description: To determine if the incidence rate of hypotensive severe/injury adverse events (IQPP DAE Classification 1.5 or 1.6) observed with the New Nomogram (Test arm) is non-inferior to the incidence rate observed with the Optimized Nomogram (Control arm).
Time Frame: From venipuncture through 72 hours post-donation.
Measure: Number; unit: Procedure with a SHAE
Units Other Than Participants: Procedures
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 3363 | 3372
Number analyzed (Procedures) | 26351 | 26117
Procedure with a SHAE | 10 | 8

7. Secondary Outcome: Time From Start of Plasmapheresis Procedure to the First SHAE
Description: To determine if the time from start of plasmapheresis procedure to the first SHAE observed with the New Nomogram (Test arm) is non-inferior to the time observed with the Optimized Nomogram (Control arm).
Time Frame: From venipuncture through end of the procedure.
Population: Procedures in which a SHAE occurred.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 44 | 42
minutes | 44.26 (10.22) | 40.53 (40.20)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from venipuncture through 72 hours post-donation. The subject had up to 2 weeks post-donation to self-report any AEs that occur through 72 hours post-donation. Adverse events were collected for the duration of the study (4 months and 23 days).
Description: For the purposes of this study, all adverse events were defined and categorized using IQPP Standard for Recording Donor Adverse Events.
  Adverse event data were monitored and assessed per procedure, rather than at the participant level.
Arm/Group | Test Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/26351 | 0/26117
Serious Adverse Events (participants affected / at risk) | 0/26351 | 0/26117
Other Adverse Events (participants affected / at risk) | 338/26351 | 309/26117
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Group (N=26351) | Control Group (N=26117)
IQPP 1.1 Hypotensive, Prefaint, No LOC (Minor) (Cardiac disorders) | 221 (221) | 201 (201)
IQPP 1.2 Hypotensive, Prefaint, No LOC (Moderate) (Cardiac disorders) | 19 (19) | 24 (24)
IQPP 1.3 Hypotensive, LOC (brief) (Cardiac disorders) | 14 (14) | 8 (8)
IQPP 1.4 Hypotensive, LOC (prolonged) (Cardiac disorders) | 1 (1) | 2 (2)
IQPP 1.5 Hypotensive, Severe (With or Without LOC) (Cardiac disorders) | 9 (9) | 8 (8)
IQPP 1.6 Hypotensive, Injury (Cardiac disorders) | 1 (1) | 0 (0)
IQPP 3. Local Injury Related to Phlebotomy (Injury, poisoning and procedural complications) | 28 (28) | 33 (33)
IQPP 4. Citrate Reaction (Blood and lymphatic system disorders) | 34 (34) | 26 (26)
IQPP 7.1 Allergic, Local (General disorders) | 3 (3) | 0 (0)
IQPP 8. Hyperventilation (General disorders) | 8 (8) | 6 (6)
IQPP 9. Other (General disorders) | 0 (0) | 1 (1) — Chest pressure/pain/tightness; unknown etiology

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The protocol, procedures, and data pertaining to this study will be treated as confidential information. Publication of data and/or information derived from these studies must be done with the prior review and approval of the Sponsor. Scientific personnel may share authorship with investigators on abstracts, oral presentations and manuscripts. The first author will be the person assuming primary responsibility for the abstract or manuscript.

DOCUMENTS (2):
  • Study Protocol (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT06122935/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT06122935/SAP_001.pdf